CLINICAL TRIAL: NCT01504789
Title: Part II: Exercise in Hispanic Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-0201; U54 (Other Grant/Funding Number: NCI); NCI-2015-01759 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2011-12-28; First posted 2012-01-05 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Cancer Survivors; Exercise; Hispanic; Mexican-American; Puerto Rican; Culturally tailored exercise; Fitness tests; Questionnaires; Surveys; Culturally tailored written material
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cultural Related Material Group (Experimental): Patients will be randomized to receive either culturally adapted AI materials or non-culturally adapted SI materials. Intervention materials will be mailed to patients every 2 weeks. Based on the results of the fitness tests, a specific exercise program will be presented. The research staff will call about every 2 weeks to check that materials were received and have been sent back whatever materials are due. The phone call should take no more than 15 minutes. At 6 months after the follow-up visit, a packet of follow-up questionnaires about physical activity and quality of life will be mailed or given over the phone. The questionnaire packet will be mailed with a postage-paid return envelope. It should take about 10 minutes to complete the questionnaires.
  Interventions: Behavioral: Baseline Fitness Test; Behavioral: Questionnaires; Behavioral: Individualized Exercise Program; Behavioral: Written Materials
- Non-Cultural Related Material Group (Experimental): Patients will be randomized to receive either culturally adapted AI materials or non-culturally adapted SI materials. Intervention materials will be mailed to patients every 2 weeks. Based on the results of the fitness tests, a specific exercise program will be presented. The research staff will call about every 2 weeks to check that materials were received and have been sent back whatever materials are due. The phone call should take no more than 15 minutes. At 6 months after the follow-up visit, a packet of follow-up questionnaires about physical activity and quality of life will be mailed or given over the phone. The questionnaire packet will be mailed with a postage-paid return envelope. It should take about 10 minutes to complete the questionnaires.
  Interventions: Behavioral: Baseline Fitness Test; Behavioral: Questionnaires; Behavioral: Individualized Exercise Program; Behavioral: Written Materials
- Waitlist Group (Active Comparator): Patients may choose to participate in the exercise program after 16-week assessment. After 4 months of exercise, all the follow-up tests repeated. Exercise recommendation then given, and all of the intervention materials.
  Interventions: Behavioral: Baseline Fitness Test; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Baseline Fitness Test — Complete fitness tests to measure strength, flexibility, balance, and aerobic capacity. All of the baseline fitness tests will be repeated at the end of the program (at about the 16th week) during a follow-up visit.
Behavioral: Questionnaires — At the baseline visit, complete questionnaires about demographic information taking about 35 minutes to complete. At 6 months after the follow-up visit, a packet of follow-up questionnaires about physical activity and quality of life will be mailed or given over the phone. It should take about 10 minutes to complete these questionnaires. Patients also be asked to fill out a questionnaire every week that asks about level of physical activity. The questionnaire should take about 5 minutes to complete.
  Other Names: Surveys
Behavioral: Individualized Exercise Program — The exercise programs will be individualized based on results from baseline fitness assessments and individual medical history using ACSM guidelines. For resistance and flexibility exercises each patient will receive an exercise prescription and instructional session prior to beginning the program. Invitation extended to attend monthly Group Exercise sessions with a family member. Resistance tubes, pedometer, exercise book, and video issued for use at home.
  Arms: Cultural Related Material Group; Non-Cultural Related Material Group
Behavioral: Written Materials — Either culturally adapted AI materials or non-culturally intervention materials will be mailed to patients every 2 weeks. The 7 themed sessions are: Getting Started;Goal Setting;Effective Energy Balance;Getting Confident;Uncovering Barriers;Lapsing, Relapsing, Collapsing;and Continuing to be Active.
  Arms: Cultural Related Material Group; Non-Cultural Related Material Group

SUMMARY:
The goal of this research study is to test an exercise program that is designed for Hispanic breast cancer survivors. Researchers want to learn the most effective strategies for promoting exercise.

DETAILED DESCRIPTION:
Study Summary:

If you are found to be eligible to take part in this study, you will come in for 2 visits to complete fitness testing and questionnaires at the Behavioral Research Treatment Center (BRTC) at MD Anderson. During the week before your first visit to the BRTC, you'll wear an accelerometer at home. An accelerometer is a small device that you wear on your waist during the day. It records how active you are. The accelerometer will be mailed to you or given to you in clinic ahead of time by a staff member. You will bring the accelerometer with you to your first visit to the BRTC. This will be repeated at the end before your follow-up assessment visit. The visits should last about 2 hours and 30 minutes. You will be asked to exercise about 3-5 times every week for 16 weeks at home for at least 30 minutes. You will also be invited to group exercise sessions every month. You should attend at least 2 of these sessions. A family member or friend is invited to attend the group sessions with you. Six (3) months after the follow-up visit, you will complete follow-up questionnaires.

Study Visits:

At the baseline (first) visit, your blood pressure, heart rate, height, and weight will be measured. Your waist and hip will be measured. A tool that measures your skin thickness will be used on the back of your arm, above your hip, and on your thigh. Your arms will be measured by placing your arm in a tool used for measuring arm volume.

You will complete questionnaires about your demographic information (such as your age), medical history, any drugs you may be taking, your current level of physical activity, your quality of life, and your environment and exercise (such as how many people you see exercising daily). The questionnaires should take about 35 minutes to complete. You may complete these questionnaires either when you sign the informed consent form or at your first visit.

Blood (about 1½ tablespoons) will be drawn during your baseline and 4-months visits after you fast (have nothing to eat or drink but water) for 12 hour. These samples will be stored for future testing on biomarkers. Biomarkers are found in the blood and may be related to breast cancer risk.

You will complete fitness tests to measure your strength, flexibility, balance, and aerobic capacity (how effectively you breathe in air while you are exercising).

For the strength tests, you will pull on a bar that is connected to a sensor that shows how much force you are using. You will pull on the bar as hard as you can for 3 seconds. You will have at least 10 seconds of rest between efforts. You will do pulls to measure the strength of your arms, shoulders, and upper body. To measure your hand and forearm muscle strength, you will squeeze and release your hand on a hand tool. To measure your leg strength, you will stand and sit back down in a chair as many times as you can in 30 seconds. You will be shown how to do each of these tests.

For flexibility, you will perform a "sit-and-reach" test and a "stand-and-reach" test. Your hip and lower back flexibility will be measured using a "sit-and-reach" flexibility box. You will sit on the floor with your feet placed on the edge of the box. You will reach forward with your hands as far as possible 3 different times. The farthest reach will measure your lower body flexibility. To measure your upper body flexibility, you will do a "stand and reach" test. You will stand next to a wall with your arm stretched forward. Then you will reach forward as far as possible without your feet lifting off the ground. The distance reached forward will be the measure of your upper body flexibility. Range of motion of your arm will be measured by asking you to lift your arm upward with your thumb pointing up. This will be done on the side and in front of you.

For aerobic testing, you will be asked to walk on a treadmill. Before you exercise, you will have an electrocardiogram (ECG) to check your heart function and your heart rate and blood pressure will be measured. A nose clip and mouthpiece will be put on you. During exercising, you will have an ECG. Your blood pressure will also be measured every few minutes. You will be asked at several times to point to a scale that measures your overall level of effort. You will walk on the treadmill at increasing speeds and inclines (hills) until you reach a point of about 85 percent of your maximum heart rate. At that point, the treadmill will be slowed down and you will be allowed to walk slowly and recover. You can ask to stop the treadmill at any time. The reason for doing this test is to see how your body reacts to hard exercise at an intensity higher than will be recommended for you during the study when you will be exercising on your own. You will be asked to perform a 6-minute walk test as a warm-up. This test measures the distance that you can walk quickly on a flat, hard surface for 6 minutes.

All of the baseline fitness tests will be repeated at the end of the program (at about the 16th week) during a follow-up visit. At the follow-up visit, you will also be asked to complete a feedback questionnaire and you will be interviewed for your feedback on the newsletters. This will help researchers design future research studies. The questionnaire and interview should take about 15 minutes to complete. You will also be asked to answer a Food Questionnaire at the follow-up visit. This questionnaire will include questions about your usual food intake during the last year. It will take about an hour to complete this questionnaire.

Study Groups:

After your baseline fitness tests and questionnaires, you will be randomly assigned (as in the flip of a coin) to 1 of 3 study groups. Groups 1 and 2 will be given an individualized exercise program, have the same amount of contact with research staff, and receive written materials about exercise. The only difference between the groups is that they will be given different written materials. Group 3 will be a "waiting list" group who choose to participate in the exercise program after their 16-week assessment. After 4 months of exercise, they will repeat all the follow-up tests described above, and receive an exercise recommendation and all the intervention materials. You will have an equal chance of being assigned to one of the three groups. You will know if you are in the waiting list group (3) or one of the exercise groups (1 or 2), but if you are in an exercise group you will not know which one.

Exercise Program:

Based on the results of the fitness tests, a specific exercise program for you will be presented to you. The comprehensive program will include aerobic (cardiovascular) training, strength training, and flexibility training to be completed at home. A set of resistance tubes will be given to you to keep and use at home. You will also be given a booklet and DVD video that contain the exercise. If you would like, after the follow-up visit, a long-term suggested exercise program will be given to you.

You will be given an exercise log to keep track of your exercising. You will also be asked to fill out a questionnaire every week that asks about your level of physical activity. The questionnaire should take about 5 minutes to complete. Every month, you will be asked to fill out a questionnaire about any swelling you may have had. This questionnaire should take about 5 minutes to complete. Every month, you will mail your completed questionnaires and exercise logs back to the study staff in postage-paid envelopes that will be provided to you.

Newsletters and Study Contact:

Every 2 weeks, you will receive a newsletter on a different theme related to exercise. One of the newsletters will be about healthy eating. The wording of the material will be different between groups, but the overall theme will be the same. The research staff will call you about every 2 weeks to check that you have received the materials and have sent back whatever materials are due. The phone call should take no more than 15 minutes. However, you can ask research staff any questions about the program at any time using the contact information that will be given to you.

Follow-up Questionnaires:

At 3 months after the follow-up visit, a packet of follow-up questionnaires about your physical activity and quality of life will be mailed to you or given over the phone. The questionnaire packet will be mailed with a postage-paid return envelope. It should take about 10 minutes to complete the questionnaires. The research staff will call you to check that you have received it and encourage you to complete it. If you are coming to MD Anderson for any appointments, you will receive the packet in person instead.

Length of Study:

Your study participation will be over after you complete the follow-up questionnaires. Your study participation may be stopped early if you become injured, if you become ineligible (for example, if you need to have treatment), or if the research staff thinks it is in your best interest.

ELIGIBILITY:
Inclusion Criteria:

1. Be Female and be 21 years of age or older. (Pilot Test and PreTest Criteria)
2. Self-reported Mexican-American ( for Mexican-American participants) or Puerto Rican ethnicity. (Pilot Test and PreTest Criteria)
3. History of breast cancer (invasive or ductal carcinoma in situ). (Pilot Test Criteria only)
4. At least 3 months post treatment (surgery, chemotherapy, radiation). (Pilot Test Criteria only)
5. Not meeting current recommended physical activity guidelines. (Pilot Test and PreTest Criteria)
6. Able to read/write in either English or Spanish. (Pilot Test and PreTest Criteria)
7. Reside in Harris County, Texas or one of the contiguous counties or metropolitan area of San Juan, Puerto Rico. (Pilot Test and PreTest Criteria)
8. Be able to provide informed consent. (Pilot Test and PreTest Criteria)
9. Be oriented to person, place, and time. (Pilot Test and PreTest Criteria)

Exclusion Criteria:

1. Currently receiving Herceptin or non-hormonal treatment for cancer (hormonal treatment is allowed). (Pilot Test and PreTest Criteria)
2. Present with any of American College of Sports Medicine's absolute contraindications to exercise testing: (A recent significant change in the resting ECG suggesting significant ischemia, recent myocardial infarction (within 2 days), or other acute cardiac event; unstable angina; uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise; symptomatic severe aortic stenosis; uncontrolled symptomatic heart failure; acute pulmonary embolus or pulmonary infarction; acute myocarditis or pericarditis; suspected or known dissecting aneurysm acute systemic infection, accompanied by fever, body aches, or swollen lymph glands). ( Pilot Test and PreTest Criteria)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in Exercise Behavior and Energy Expenditure | 6 months
  Exercise behavior measured as frequency of exercise as assessed by the IPAQ score. Multiple linear regression used to test for differences in the changes between groups adjusting for relevant covariates, such as baseline activity level (IPAQ score) and BMI. Linear mixed model analysis also performed for weekly change in exercise behavior. The continuous score (MET minutes/week) used as primary physical activity outcome, measured at baseline and follow-up. Compliance measured using exercise logs, which will record resistance exercise and pedometer steps.

SECONDARY OUTCOMES:
Effects of Behavioral Exercise Intervention on Biological Markers | 16 weeks
  Blood (about 1½ tablespoons) collected at baseline and 4 months visits following a 12-hour fast. Blood will be processed and stored for later biomarker analysis - body adiposity, sex hormone binding globulin, estradiol, adipokines (adiponectin, leptin, resistin), cytokines (TNF, CRP, IL-6).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PHD, BA, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Palacios C, Daniel CR, Tirado-Gomez M, Gonzalez-Mercado V, Vallejo L, Lozada J, Ortiz A, Hughes DC, Basen-Engquist K. Dietary Patterns in Puerto Rican and Mexican-American Breast Cancer Survivors: A Pilot Study. J Immigr Minor Health. 2017 Apr;19(2):341-348. doi: 10.1007/s10903-016-0398-y. PMID 26984227
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org